CLINICAL TRIAL: NCT01616056
Title: A Single Center Phase II Study of Bandage Lenses for Ocular Graft-Versus-Host Disease After Allogeneic Hematopoietic Cell Transplantation
Brief Title: Bandage Lenses in Treating Patients With Ocular Graft-Versus-Host Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Stephanie Lee, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2617.00; NCI-2012-00862 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2617.00 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2012-06-06; First posted 2012-06-11 (Estimated); Results first posted 2017-07-17 (Actual); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Graft Versus Host Disease; Ophthalmologic Complications
Keywords: Chronic graft-versus-host disease; eye
MeSH Terms: conditions — Graft vs Host Disease; Bronchiolitis Obliterans Syndrome | interventions — Therapeutics; Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bandage Contact Lenses (Experimental): Patients wear bandage lenses continuously for at least 3 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: graft versus host disease prophylaxis/therapy; Other: questionnaire administration; Procedure: optical coherence tomography

INTERVENTIONS:
Biological: graft versus host disease prophylaxis/therapy — Wear bandage lenses
  Other Names: prophylaxis/therapy, graft versus host disease; prophylaxis/therapy, GVHD
Other: questionnaire administration — Ancillary studies
Procedure: optical coherence tomography — Optional ancillary studies

SUMMARY:
This phase II clinical trial studies how well bandage lenses work in treating patients with ocular graft versus host disease. Bandage lenses may be helpful in relieving eye symptoms and damage caused by eye graft versus host disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the symptom improvement after 2 weeks of therapy with bandage lenses.

SECONDARY OBJECTIVES:

I. To confirm short-term safety within 1 month after bandage lenses.

II. To determine improvement in ophthalmologic examinations after bandage lenses.

III. To explore the use of optical coherence tomography as an objective measure of corneal inflammation.

OUTLINE:

Patients wear bandage lenses continuously for at least 3 months in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic graft versus host disease (GVHD) as defined by the National Institutes of Health (NIH) criteria
* Ocular symptoms of NIH eye score 2 or greater:

  * Score 2: Moderate dry eye symptoms partially affecting activities of daily living (ADL) (requiring drops > 3 x per day or punctal plugs), WITHOUT vision impairment
  * Score 3: Severe dry eye symptoms significantly affecting ADL (special eyewear to relieve pain) OR unable to work because of ocular symptoms OR loss of vision caused by keratoconjunctivitis
* No new systemic immunosuppressive medications within 1 month prior to enrollment
* Subject has the ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* Absolute neutrophil count < 1000/ul
* Known hypersensitivity or allergy to contact lenses
* Evidence of any active viral, bacterial, or fungal infection in the eyes that is progressive despite appropriate treatment
* Treatment with contact lenses within the previous 3 months for any indication
* Active psychiatric disorder, substance abuse or any other reason that would interfere with compliance with the study protocol

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-06; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Lee, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
All data are available now for sharing. Researchers must contact Stephanie Lee and sign a data use agreement.

REFERENCES:
- [Result] Inamoto Y, Sun YC, Flowers ME, Carpenter PA, Martin PJ, Li P, Wang R, Chai X, Storer BE, Shen TT, Lee SJ. Bandage Soft Contact Lenses for Ocular Graft-versus-Host Disease. Biol Blood Marrow Transplant. 2015 Nov;21(11):2002-7. doi: 10.1016/j.bbmt.2015.07.013. Epub 2015 Jul 17. PMID 26189353

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bandage Contact Lenses
Started | 20
Completed | 19
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Bandage Contact Lenses
Number analyzed (Participants) | 19
Age, Continuous [Median (Full Range); unit: years] | 55 [32 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 15
  More than one race | 1
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Patient-reported Symptoms Measured by the 8-point Lee Eye Subscale
Description: Lee eye subscale: sx6 dry eyes, sx7 need to use eye drops frequently, sx8 difficulty seeing clearly 0=not at all, 4=extremely bothered. If have at least one of (sx6,sx7,sx8), then sx_eye=mean(sx6,sx7,sx8)*25. Minimum possible score: 0 correlated with better outcome, maximum score possible: 100 correlated with worse outcome. Clinically meaningful change is half a standard deviation, which is a decrease of 11.8 of more for this scale.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bandage Contact Lenses
Number analyzed (Participants) | 19
units on a scale
  Baseline | 75.4 (4.25)
  2 weeks | 63.2 (4.82)
  4 weeks | 61.8 (4.52)
  3 months | 56.3 (7.28)
Statistical Analysis 1: Comparison: Bandage Contact Lenses; Test type: Superiority; p = 0.01, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Number of Participants Who Perceived a Clinically Meaningful Change as Measured by the 8-level Lee Eye Symptom Subscale
Description: 8-level change score is from 0 completely gone to 7 very much worse. Clinically meaningful improvement is defined as half a standard deviation (decreased score of 11.8 or greater).
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Bandage Contact Lenses
Number analyzed (Participants) | 19
Participants
  2 weeks | 9
  4 weeks | 11
  3 months | 9

3. Primary Outcome: Change in Patient-reported Symptoms as Measured by the Ocular Surface Disease Index
Description: OSDI minimum score: 0, correlated with better outcome, maximum score: 100, correlated with worse outcome. 12 questions 0 none of the time to 4 all of the time. (Sum of scores)x25/number of questions answered. Clinically meaningful change scores are half a standard deviation, which is 10.9 for the OSDI.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bandage Contact Lenses
Number analyzed (Participants) | 19
units on a scale
  Baseline | 54.5 (6.19)
  2 weeks | 36.8 (5.32)
  4 weeks | 32.9 (5.74)
  3 months | 35.6 (6.50)
Statistical Analysis 1: Comparison: Bandage Contact Lenses; Test type: Superiority; p = 0.002, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Number of Participants Who Perceived a Clinically Meaningful Change as Measured by the OSDI
Description: as for outcome 3
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Bandage Contact Lenses
Number analyzed (Participants) | 19
Participants
  2 weeks | 10
  4 weeks | 13
  3 months | 10

5. Primary Outcome: Change in Patient-reported Symptoms as Measured by the 11-point Eye Rating Scale
Description: The 11-point eye scale goes from 0 not present to 10 as bad as you can imagine. Clinically meaningful change is defined as a 2 point or more decrease.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bandage Contact Lenses
Number analyzed (Participants) | 19
units on a scale
  Baseline | 7.11 (0.42)
  2 weeks | 5.00 (0.56)
  4 weeks | 4.37 (0.45)
  3 months | 3.94 (0.59)
Statistical Analysis 1: Comparison: Bandage Contact Lenses; Test type: Superiority; p = 0.001, Wilcoxon (Mann-Whitney)

6. Primary Outcome: Number of Participants Who Perceived a Clinically Meaningful Change as Measured by the 11-point Eye Scale
Description: as for outcome 5
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Bandage Contact Lenses
Number analyzed (Participants) | 19
Participants
  2 weeks | 11
  4 weeks | 13
  3 months | 12

7. Secondary Outcome: Number of Patients Who Experienced Serious Adverse Events
Description: Safety of Bandage Contact Lenses at 1 month
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Bandage Contact Lenses
Number analyzed (Participants) | 19
Participants | 0

8. Secondary Outcome: Change in Comprehensive Ophthalmologic Evaluations
Description: LogMAR visual acuity score of 0 is equivalent to 20/20 vision. Patients were assessed by ophthalmologists at enrollment, 2 weeks and afterwards as medical needed.
Time Frame: 2 weeks
Population: Ophthalmology assessments made after 2 weeks were not analyzed because of incomplete data collection.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Bandage Contact Lenses
Number analyzed (Participants) | 19
logMAR
  logMAR visual acuity baseline | 0.26 (0.030)
  logMAR visual acuity 2 weeks | 0.15 (0.030)
Statistical Analysis 1: Comparison: Bandage Contact Lenses; Test type: Superiority; p = 0.005, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Change in Optical Coherence Tomography
Description: Patients were assessed by ophthalmologists at enrollment, 2 weeks and afterwards as medical needed.
Time Frame: 2 weeks
Population: Optical coherence tomography results were not analyzed because of incomplete data collection.
Arm/Group | Bandage Contact Lenses
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Bandage Contact Lenses
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 14/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bandage Contact Lenses (N=19)
Foreign body sensation (Eye disorders) | 14 (14)
Swollen eye lids (Eye disorders) | 5 (5)
Excessive tearing (Eye disorders) | 2 (2)
Corneal edema and stromal haze (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No